CLINICAL TRIAL: NCT06043128
Title: The Relatıonshıp Of Proprıoceptıve Awareness Wıth Balance And Spastıcıty In Patıents Wıth Stroke Wıth Dıfferent Trunk Impact Levels
Brief Title: Proprioceptive Awareness in Stroke Patients With Different Trunk Impact Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Güler ERTUĞRUL, MSc student, physiotherapist, Suleyman Demirel University
Other Study IDs: 573
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Stroke; Balance; Proprioception; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with High Body Control: This group consists of stroke patients who received 23 or close to 23 points on the trunk impairment scale. In these patients, muscle stiffness, awareness of the sense of balance and position, quality of life will be evaluated and their relationships will be examined.
  Interventions: Other: Patients With Stroke With Different Trunk Impact Levels
- Group with Low Body Control: This group consists of stroke patients who received 0 points or close to 0 points from the trunk impairment scale. In these patients, muscle stiffness, awareness of the sense of balance and position, quality of life will be evaluated and their relationships will be examined.
  Interventions: Other: Patients With Stroke With Different Trunk Impact Levels

INTERVENTIONS:
Other: Patients With Stroke With Different Trunk Impact Levels — Before the study, written and verbal "Informed Consent Form" will be obtained from all participants who meet the inclusion criteria.Trunk Impairment Scale (TRS) will be used to measure trunk control, which is our independent variable. Scores close to 23 points on the TIS will constitute the group with high trunk control, and those with scores close to 0 will constitute the group with low trunk control. Spasticity of the participants, Modified Tardiue Scale (MTS), cervical proprioceptive awareness cervical joint error test, lower extremity proprioceptive awareness Proprioception test in Technobody Prokin 252 Isokinetic Balance Platform, balance skills Dynamic and static balance in Tecnobody Prokin 252 Isonkinetic Balance Platform will be evaluated by tests. The patients' quality of life will be evaluated with the stroke-specific quality of life scale. All data obtained will be noted on a prepared evaluation form.
  Other Names: Group with Low Body Control; Group with High Body Control

SUMMARY:
Trunk control is important for maintaining an upright posture, increasing the quality of movement during dynamic activities, and performing transfer activities safely. Individuals with stroke, which is one of the most common neurological diseases in the world, may have various degrees of trunk affect because the contraction strength of the trunk muscles and their ability to work in harmony with each other are reduced. Depending on the increase in the level of trunk involvement, proprioceptive deterioration, increase in balance problems and deterioration in spasticity characteristics can be observed in patients. However, the relationship between these disorders in individuals with stroke, independent of trunk involvement, has not been defined. Therefore, in this study, we aimed to examine the relationship between proprioceptive awareness and balance and spasticity in stroke patients with different trunk involvement levels. 98 chronic stroke patients will be included in the study. Before the study, written and verbal "Informed Consent Form" will be obtained from all participants who meet the inclusion criteria. After recording the sociodemographic and clinical characteristics of the participants, the cognitive status of the patients will be evaluated with a mini mental test. Trunk Impairment Scale (TRS) will be used to measure trunk control, which is our independent variable. GBS will be administered by another physiotherapist who is blinded to the study. Participants will be divided into two groups, high and low trunk control, according to the score obtained from the GBS. Spasticity of the participants, Modified Tardiue Scale (MTS), cervical proprioceptive awareness cervical joint error test, lower extremity proprioceptive awareness Proprioception test in Technobody Prokin 252 Isokinetic Balance Platform, balance skills Dynamic and static balance in Tecnobody Prokin 252 Isonkinetic Balance Platform will be evaluated by tests. The patients' quality of life will be evaluated with the stroke-specific quality of life scale. In order to prevent bias, scores obtained from the GBÖ will not be shared with the physiotherapist who performs other tests. All data obtained will be noted on a prepared evaluation form. After all data is collected, intra-group and inter-group comparisons will be made.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 98 chronic stroke patients will be included in the study. Written and verbal "Informed Consent Form" will be obtained from all participants who meet the inclusion criteria for the study. After the sociodemographic and clinical characteristics of the participants are recorded, the cognitive status of the patients will be evaluated with a mini mental test. The Trunk Disability Scale (TRS) will be used to measure trunk control, which is our independent variable. GBS will be administered by another physiotherapist who is blinded to the study. Participants will be divided into two groups, high and low trunk control, according to the score they receive from the GBÖ. Scores close to 23 points on the GBS will constitute the group with high trunk control, and those with scores close to 0 will constitute the group with low trunk control. The spasticity of the participants will be evaluated with the Modified Tardiue Scale (MTS), the spasticity of the muscles, and the proprioceptive awareness of the cervical region with the cervical joint error test. Lower extremity proprioceptive awareness will be evaluated with proprioception testing on the Technobody Prokin 252 Isokinetic Balance Platform, and balance skills will be evaluated with dynamic and static balance tests on the Tecnobody Prokin 252 Isonkinetic Balance Platform. The patients' quality of life will be evaluated with a stroke-specific quality of life scale. In order to prevent bias, scores obtained from the GBÖ will not be shared with the physiotherapist performing other tests. All data obtained will be noted on the prepared evaluation form. After all data is collected, intra-group and inter-group comparisons will be made.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 35-65
* Being diagnosed with stroke
* Having a stroke for the first time
* Mini Mental Test (MMT) Score ≥ 24
* Brunnstorm lower extremity stage ≥ 4
* Being clinically stable

Exclusion Criteria:

* Mini Mental Score <24 points
* Having cervical pain of 5 or higher on the visual analog scale
* Having serious vestibular, auditory and visual problems that affect balance (vertigo, etc.)
* Having a history of orthopedic surgery for the trunk and lower extremities
* Presence of an additional neurological disease (MS, Parkinson, Alzheimer's)
* Having joint rigidity that will prevent proprioceptive evaluation

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will consist of stroke patients who live in Kocaeli province and exhibit a hemiplegic-hemiparetic picture for at least 6 months after the stroke event.
Sampling Method: Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Trunk impairment scale | 20 minutes
  It consists of 3 items with different scoring alternatives. The dynamic sitting balance subscale consists of 10 items with 0 and 1 scoring options. The coordination subscale includes 4 items with different scoring alternatives. Possible compensatory strategies used during the administration of Trunk impairment scale to the patient are also evaluated. After all items have been evaluated 3 times, the best result is recorded as the patient's performance value. A score of 23 from the scale indicates that optimal trunk control is achieved, while a score approaching 0 indicates that trunk control has decreased. Turkish validity and reliability study of Trunk impairment scale in stroke patients Sag et al. Made by.
Modified Tardieu Scale | 25 minutes
  Modified Tardieu Scale consists of parameters that evaluate the angle and degree of spasticity. The scale evaluates spasticity at three different speeds in order to evaluate the speed-dependent effect of spasticity. These velocities are defined as V1, V2 and V3 velocities. V1 speed represents the evaluation at the lowest speed and V3 represents the evaluation at the highest speed. In all 3 speeds, the target joints are moved passively within the full range of motion, and the value range at which spasticity is observed is calculated by the goniometer. Spasticity degree is made between 0-4. "0" indicates no spasticity, "4" indicates indefatigable clonus (>10 seconds while mainta)
Evaluation of Proprioceptive Awareness | 30 minutes
  Cervical Joint Position Error Test will be applied to evaluate the awareness of the sense that detects neck position. Patients are seated in a chair with back support, 90 cm away from the target board fixed to the wall. Patients are first asked to memorize the position without their head tilting in any direction and try to find the same point after an active head movement. Active head movements include flexion, extension, and right and left rotations. The desired movements are repeated 10 times. After the movement, the horizontal, vertical and global distances of each point returned to the starting point will be recorded. To calculate the test result, the average values of the incorrect distances in centimeters will be calculated.
Evaluation of static and dynamic balance | 15 minutes
  To measure balance performance, patients are given a movable balance platform on the Tecnobody Prokin 252 balance platform, powered by air piston servo motors. The patient is raised on the platform that detects the sensitive measurement, which can be both movable and fixed. Thanks to the automatic engine locking function, the system instantly switches from dynamic to static measurement and provides measurement of two different balances with objective results.
Stroke-Specific Quality of Life Scale | 10 minutes
  It consists of 12 subsections, including energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision and work efficiency, and a total of 49 items. In PESS, increasing the total score indicates that the quality of life increases, while decreasing the total score indicates that the quality of life decreases.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLER ERTUĞRUL, Principal Investigator — Süleyman Demirel University Faculty of Health Sciences; MEHMET DURAY, Study Director — Süleyman Demirel University Faculty of Health Sciences
Locations (1):
- Güler Ertuğrul, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No